CLINICAL TRIAL: NCT07220161
Title: Innovative Repurposing of Trigeminal Nerve Stimulation of the Treatment of Epilepsy in Veterans
Brief Title: Trigeminal Nerve Stimulation of the Treatment of Epilepsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Hina Dave, Principal Investigator, Baylor College of Medicine
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-55827
Record Dates: First submitted 2025-10-21; First posted 2025-10-23 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Epilepsy (Treatment Refractory)
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Intervention Model Description: Cefaly Connected
Masking Description: There are no parties who are masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment with Trigeminal Nerve Stimulation (Experimental): Treatment with trigeminal nerve stimulation x 6 months
  Interventions: Device: Trigeminal nerve stimulation
- Control (No Intervention): Standard care x 6 months

INTERVENTIONS:
Device: Trigeminal nerve stimulation — The study device, "Cefaly® Connected", is a non-invasive neuromodulation tool designed for the prevention and treatment of migraine headaches. It works by delivering transcutaneous electrical stimulation to the bilateral supraorbital nerves, which are branches of the trigeminal nerve. The device is placed on the forehead, and it emits electrical impulses that modulate the activity of the trigeminal nerve.
  Arms: Treatment with Trigeminal Nerve Stimulation

SUMMARY:
Background: Epilepsy is a common neurological disorder among veterans. Medications do not control seizures in 1/3rd of patients, who often require neurostimulation. However, current neurostimulation devices are invasive. Objective: The investigators propose a novel clinical trial to repurpose the FDA-approved Cefaly device, designed for migraine relief, to treat epilepsy. The Cefaly device works by non-invasive Trigeminal neurostimulation (TNS). TNS has previously shown promising preliminary results in seizure improvement. Design: The investigators will engage 24 veterans with drug-resistant epilepsy, half of whom will receive standard care, while the other half will receive standard care plus Cefaly. This will be followed by a crossover of the treatment/control groups. The primary objective is to evaluate seizure frequency improvement over 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 65 years of age at time of consent
* Subject must have a confirmed diagnosis of epilepsy of at least 1 year, specified as focal onset epilepsy.
* Focal epilepsy with motor signs
* A minimum seizure frequency of one seizure over a 4-week period
* Subject must have failed to achieve seizure control with at least two appropriate antiseizure medications (ASM) based on the 2009 ILAE definition of drug resistant epilepsy
* Current treatment with at least 1 ASM with stable doses for at least three months

Exclusion Criteria:

* Any condition that would impact a subject's ability to follow study procedures or subject's safety
* History of significant adverse reactions to electrical stimulation (e.g. TEMS device)
* Subjects with only focal aware nonmotor seizures
* Women of childbearing age, pregnant or breastfeeding
* Implanted cardiac pacemaker or implanted/wearable defibrillator or implanted metallic device in head

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2026-05-08 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Seizure frequency | 6 months
  The primary outcome will be the reduction in seizure frequency with the treatment device compared to baseline measurements.

SECONDARY OUTCOMES:
QOLIE-31 | 6 months
  Improvement in quality of life as a secondary outcome with a focus on daily functionality, mental health, and overall subject well-being. This will be collected through the QOLIE-31.
Beck Depression Inventory | 6 months
  Mood will be followed with the Beck Depression Inventory.

CONTACTS AND LOCATIONS:
Overall Officials: Hina Dave, MD, Principal Investigator — Baylor College of Medicine/Debakey VA Medical Center
Locations (1):
- Debakey VA Medical Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magis D, Sava S, d'Elia TS, Baschi R, Schoenen J. Safety and patients' satisfaction of transcutaneous supraorbital neurostimulation (tSNS) with the Cefaly(R) device in headache treatment: a survey of 2,313 headache sufferers in the general population. J Headache Pain. 2013 Dec 1;14(1):95. doi: 10.1186/1129-2377-14-95. PMID 24289825